CLINICAL TRIAL: NCT00001547
Title: A Magnetic Resonance Spectroscopy Study of Neuropsychiatric Effects Associated With Cytokines
Brief Title: Neuropsychiatric Effects of Interferon-Alpha and Ribavirin
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960103; 96-M-0103
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Mental Disorder
Keywords: Drug; Imaging; Brain; Metabolism; Organic Mental Syndrome; Magnetic Resonance Imaging; Spectroscopy; Neuropsychiatric Disorders; Drug Effects; Interferon-alpha
MeSH Terms: conditions — Mental Disorders

SUMMARY:
Use of the drug interferon-alpha (IFN-A), is associated with frequent and well characterized side effects like neurotoxicity. Neurotoxicity can cause symptoms of depression, agitation, anxiety, and/or confusion.

The NIDDK is conducting a research study called, "Combination of Alpha Interferon with Long Term Ribavirin Therapy for Patients with Chronic Hepatitis C" (98-DK-0003). Patients participating in it are receiving interferon-alpha in addition to an antiviral medication called ribavirin. Researchers at the NIMH intend to study patients to learn more about how different medications can influence mood, thoughts and behavior.

The primary purpose of this study is to determine if treatment with IFN-A in combination with ribavirin alters human brain biochemistry as measured by proton magnetic resonance spectroscopy (MRS).

MRS uses strong magnetic fields in order to measure biochemical products of metabolism found in the brain. Researchers intend to perform MRS scans before, during, and after patients receive their medications

Researchers believe that the combination of IFN-A/Ribavirin will directly affect specific areas of the brain and as a result, some patients will develop specific mood or cognitive symptoms. Patients often must stop taking these medications because of the side effects.

This study will not contribute directly to the treatment of patient's Hepatitis C condition. However, the information gathered from this study will help researchers better understand the neuropsychiatric affects associated with interferon alpha and ribavirin therapy.

DETAILED DESCRIPTION:
The systemic administration of interferon-alpha (IFN-A) is associated with frequent and well characterized neuropsychiatric toxicity. The primary purpose of this study is to determine if treatment with IFN-A in combination with ribavirin alters human brain biochemistry as measured by proton magnetic resonance spectroscopy. The study population will be drawn from subjects simultaneously enrolled in a NIDDK protocol (98-DK-0003) that employs IFN-A and ribavirin for the treatment of hepatitis C virus (HCV) infection. Subjects will be evaluated prior to IFN-A/ribavirin treatment and then followed prospectively with the specific aim of identifying the emergence of central nervous system (CNS) effects. The principal outcome measures will be as follows: determinations of specific brain metabolites as measured by proton magnetic resonance spectroscopy (1H-MRS), a brief, non-invasive, and minimal risk procedure; ratings of mood, cognitive, and behavioral symptoms.

The hypotheses being tested in this study are as follows:

1. Treatment with IFN-A/ribavirin will decrease measures of neuronal integrity (NAA/CRE ratio) in a brain region specific fashion.
2. The degree of change in NAA/CRE in certain brain regions (e.g. prefrontal cortex) will correspond to the development of mood or cognitive symptoms.

The questions being asked in this study are relevant to the clinical management of HCV patients, since adverse neuropsychiatric effects of IFN-A and ribavirin frequently complicate protocol participation and occasionally result in a subject being taken off protocol. There are no anticipated number of patient days per year required for this study, as all participants will be simultaneously enrolled in NIDDK protocol 98-DK-0003.

ELIGIBILITY:
Subjects must be at least 18 years of age.

Subjects eligible for this study will be those enrolled in NIDDK protocol 98-DK-0003 and consequently at increased risk for the development of neuropsychiatric toxicity.

Subjects must be able to provide informed consent.

No individuals who are critically ill or markedly agitated or confused.

No individuals with implanted cardiac pacemakers or autodefibrillators.

No individuals with implanted neural pacemakers.

No individuals with CNS aneurysmal clips.

No individuals with cochlear implants.

No individuals with metallic foreign bodies in the eye or CNS.

No individuals with any form of implanted wire or metal device which may concentrate radiofrequency fields.

No pregnant women.

No individuals with a history of moderate to severe claustrophobia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1996-06; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Trzepacz PT. The neuropathogenesis of delirium. A need to focus our research. Psychosomatics. 1994 Jul-Aug;35(4):374-91. doi: 10.1016/S0033-3182(94)71759-X. PMID 7916159
- [Background] Dager SR, Steen RG. Applications of magnetic resonance spectroscopy to the investigation of neuropsychiatric disorders. Neuropsychopharmacology. 1992 Jun;6(4):249-66. PMID 1632893
- [Background] Ross BD, Jacobson S, Villamil F, Korula J, Kreis R, Ernst T, Shonk T, Moats RA. Subclinical hepatic encephalopathy: proton MR spectroscopic abnormalities. Radiology. 1994 Nov;193(2):457-63. doi: 10.1148/radiology.193.2.7972763.